CLINICAL TRIAL: NCT07070310
Title: DELirium, Incidence, preVEntion and pRogression During Acute Intensive Neurological -Neurosurgical Rehabilitation (Delirinzidenz Und Verlauf während Des Aufenthaltes in Der Neurologisch- Neurochirurgischen Frührehablilitation Der Phase B (NNFR))
Brief Title: DELirium, Incidence, preVEntion and pRogression During Acute Intensive Neurological -Neurosurgical Rehabilitation
Acronym: DeliVeriNN
Status: Not yet recruiting | Type: Observational
Sponsor: Heart Centre Rotenburg (Other)
Responsible Party: Principal Investigator, Ralf Degenhardt, PhD, Head of Clinical Research Institute, Heart Centre Rotenburg
Other Study IDs: DeliVeriNN-01
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Neurological Conditions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this longitudinal cohort study the incidence of delirium is assessed for all patients being admitted to the acute intensive neurological-neurosurgical rehabilitation over 3 years. Delirium assessment will be performed daily from admission to discharge. Patients will be divided into 3 groups, according to the presentation of delirium on admission, during the course or not any during the stay in acute rehabilitation and compared regarding the treatment and outcome.

ELIGIBILITY:
Inclusion Criteria:

* Any patient admitted to acute neurological-seurosurgical rehabilitation

Exclusion Criteria:

* : patients with level of consciousness of coma or vegetative state

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in Neurosurgical rehabilitation
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2028-08-15 (Estimated); Study Completion 2029-02-15 (Estimated)

PRIMARY OUTCOMES:
incidence of delirium | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Herz-Kreislauf-Zentrum Klinikum Hersfeld Rotenburg GmbH, Klinik für Neurologie und Neurologische Rehabilitation, Rotenburg an der Fulda, Germany

IPD SHARING:
Plan to Share IPD: No